CLINICAL TRIAL: NCT04736420
Title: Replication of the EINSTEIN-DVT Anticoagulant Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-EINSTEIN-DVT
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Warfarin: Reference group
  Interventions: Drug: Warfarin
- Rivaroxaban: Exposure group
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban dispensing claim is used as the exposure group
  Groups: Rivaroxaban
Drug: Warfarin — Warfarin dispensing claim is used as the reference group
  Groups: Warfarin

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates through standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Criteria:

Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Inclusion Criteria:

- Confirmed acute symptomatic proximal DVT without symptomatic PE

Exclusion Criteria:

* Age ≤ 18
* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of DVT or PE two weeks prior to and including day of enrollment
* Other indications for VKA than DVT and/or PE six months prior to and including day of enrollment
* Any of the following six months prior to and including day of enrollment:

  * Creatine clearance < 30 ml/min
  * Significant liver disease (e.g. acute hepatitis, chronic active hepatitis, cirrhosis) or ALAT>3 ULN
  * Bacterial endocarditis
  * Active bleeding or high risk for bleeding contraindicating treatment with enoxaparin or VKA
  * Systolic blood pressure > 180 mgHg or diastolic blood pressure > 110 mgHg
  * Childbearing potential without proper contraceptive measures, pregnancy, or breastfeeding
* Life expectancy < 3 months in the last year prior to and including day of enrollment
* Concomitant use of strong CYP3A4 inhibitors (e.g. HIV protease inhibitors, systemic ketoconazole) or strong CYP3A4 inducers two weeks prior to and including day of enrollment
* Symptomatic pulmonary embolism two weeks prior to and including day of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing rivaroxaban to warfarin users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of rivaroxaban or warfarin (index date). We will restrict the analyses to patients with a diagnosis of proximal DVT without symptomatic PE.
Sampling Method: Non-Probability Sample
Enrollment: 78605 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of venous thromboembolism | Through study completion or point of censoring, up to 12 months
  Claims-based algorithm: see attached protocol for full definition

SECONDARY OUTCOMES:
Relative hazard of a major bleeding event | Through study completion or point of censoring, up to 12 months
  Claims-based algorithm: see attached protocol for full definition

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT04736420/Prot_SAP_001.pdf